CLINICAL TRIAL: NCT02319213
Title: The Increase of Intra-abdominal Pressure Can Affect Intra-ocular Pressure.
Brief Title: This Study Performed to Develop a New Technique for Measuring the Intra Abdominal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, İlhan Ece, Department of Surgery., Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SU 08-38
Record Dates: First submitted 2014-12-07; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Abdominal Compartment Syndrome
Keywords: Intra-abdominal pressure,; intraocular pressure,; abdominal hypertension,; laparoscopy,; critical care
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group C (No Intervention): The control group (Group C) was not subjected to laparoscopic intervention
- Group L (Experimental): Intraocular pressure measurement with 9 mmHg insufflation
  Interventions: Other: Intraocular pressure measurement with 9 mmHg insufflation
- Group M (Experimental): Intraocular pressure measurement with 12 mmHg insufflation
  Interventions: Other: Intraocular pressure measurement with 12 mmHg insufflation
- Group H (Experimental): Intraocular pressure measurement with 15 mmHg insufflation
  Interventions: Other: Intraocular pressure measurement with 15 mmHg insufflation

INTERVENTIONS:
Other: Intraocular pressure measurement with 9 mmHg insufflation — Comparison of intraocular pressure levels at different abdominal pressure
  Arms: Group L
Other: Intraocular pressure measurement with 12 mmHg insufflation — Comparison of intraocular pressure levels at different abdominal pressure
  Arms: Group M
Other: Intraocular pressure measurement with 15 mmHg insufflation — Comparison of intraocular pressure levels at different abdominal pressure
  Arms: Group H

SUMMARY:
The purpose of this study is to evaluate the changes of intraocular pressure due to the increase of intra abdominal pressure.

DETAILED DESCRIPTION:
In this prospective study, 40 patients undergoing elective surgery were included. Patients were divided into four groups of 10 patients. The control group (Group C) was not subjected to laparoscopic intervention. Laparoscopic surgery was respectively performed with an intra-abdominal pressure of 9, 12 and 15 mmHg in Groups L (low), M (medium), and H (high pressure). Intraocular pressure was measured binocularly in each patient at three different time (before, during and end of surgery) using a contact tonometer.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 30 kg/m2 or less
* American Society of Anesthesiologists (ASA) status I-II

Exclusion Criteria:

* Pre-existing eye disease,
* Cardiovascular or neuromuscular disease,
* Difficult intubation,
* The use of any antihypertensive agents.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
intra-abdominal pressure | 1 day after the surgery.
  Changes in intraabdominal pressure

CONTACTS AND LOCATIONS:
Overall Officials: İlhan Ece, Study Director — Selcuk Universitesi Tip Fakultesi Genel Cerrahi poliklinigi
Locations (1):
- Selcuk University, Konya, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Ece I, Vatansev C, Kucukkartallar T, Tekin A, Kartal A, Okka M. The increase of intra-abdominal pressure can affect intraocular pressure. Biomed Res Int. 2015;2015:986895. doi: 10.1155/2015/986895. Epub 2015 Jan 14. PMID 25648230